CLINICAL TRIAL: NCT05024643
Title: Outcome of the Endoscopic Repair of Frontal Sinus Cerebrospinal Fluid Leak
Brief Title: Endoscopic Repair of Frontal Sinus CSF Leak
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdulkarim Hasan, Laboratory manager, Al-Azhar University
Other Study IDs: 21-01-010
Record Dates: First submitted 2021-08-22; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: CSF Leakage
MeSH Terms: conditions — Cerebrospinal Fluid Rhinorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endonasal endoscopy — Complete sphenoethmoidectomy; Draf type IIa, IIb, and III according to defect location.
  Defect less than 3 mm closed by a plug of fat and facia lata or middle turbinate mucosa.
  Defect more than 3 mm closed by underlying facia lata, underlying cartilage, and overlay facia lata.

SUMMARY:
This retrospective study was conducted on patients with frontal sinus leaks came to ENT departments of Al-Azhar University Hospital, New Damietta, Egypt, for a period of five years.

DETAILED DESCRIPTION:
All patients in this study were evaluated during the follow-up period. Patients' age, sex, occupation, residence, and telephone number were recorded for each participant for demographic purposes. General and local examinations were also performed preoperatively as usual.

Medical history, surgical approach, leakage site, complications, reconstruction technique, and follow-up were recorded.

All cases were treated by endonasal endoscopy

* Complete sphenoethmoidectomy.
* Draf type IIa, IIb, and III according to defect location.
* Defect less than 3 mm closed by a plug of fat and facia lata or middle turbinate mucosa.
* Defect more than 3 mm closed by underlying facia lata, underlying cartilage, and overlay facia lata.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent endoscopic frontal sinus repair. Traumatic or spontaneous patients with a CSF leak at a minimum of six months not responding to conservative measures were included.

Exclusion Criteria:

* Known malignancy or patients with frontal leak due to extensive tumor resection or intracranial injury

Ages: 10 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with frontal sinus leaks attended Al-Azhar University Hospital, New Damietta, Egypt
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Successful treatment | 1 year
  Intracranial tension from 7-15 mmHg, No leakage, No complications

SECONDARY OUTCOMES:
Complications | 1 week
  Elevated intracranial tension, more than 15 mmHg, Fever, more than 37.5 degree, Meningitis

IPD SHARING:
Plan to Share IPD: Undecided